CLINICAL TRIAL: NCT07243548
Title: Effect of Peripheral Magnetic Stimulation in Patients With Chronic Lower Back Pain - Controlled, Randomized Clinical Trial
Brief Title: Effect of Peripheral Magnetic Stimulation in Patients With Chronic Lower Back Pain
Acronym: PEMS-CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Principal Investigator, Inês Gomes, Research Support Office, Egas Moniz - Cooperativa de Ensino Superior, CRL
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEEM1329
Record Dates: First submitted 2025-04-16; First posted 2025-11-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain
Keywords: Peripheral magnetic stimulation; low back pain; chronic pain; neuromodulation
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Individuals with chronic low back pain with a score between 40 and 80 on the Oswestry scale will be selected, and 50 will be selected for treatment at the Physiotherapy School of the Federal University of Alfenas - MG and the Egas Moniz University Clinic - CUEM. The individuals will be divided into 2 groups: the control group and the intervention group.
  The volunteers will be divided into a control group and an intervention group through randomization. To this end, the participants will be allocated by another researcher, who will use the Research Randomizer website into two groups: Control Group (CG) and Intervention Group (IG).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rPMS Controle (Experimental): For patients in the rPMS control group, also in the prone position, the coil will be applied in a transverse orientation to the most painful lumbar region. This position of the coil, at a 90° angle to the body surface, will minimize the effects of the magnetic stimulation applied to the area.
  Interventions: Device: rPMS Controle
- rPMS Intervention (Experimental): For patients in the rPMS intervention group - in the prone position - the coil will be placed in a flat tangential orientation targeting the most painful lumbar region. This will allow the coil to be positioned parallel to the body surface, thus maximizing the effects of the magnetic stimulation applied to the area.
  Interventions: Device: rPMS Intervention

INTERVENTIONS:
Device: rPMS Intervention — Both groups will undergo 10 sessions over a 2-week period. Each session will last 20 minutes and will be intermittent stimulation protocol consisting of 5 seconds of stimulation at a frequency of 20 Hz followed by 25 seconds of rest. The total number of stimulations over 20 minutes will be 4,000 pulses.
  The stimulation intensity level will be set at the level that induces sufficient contraction of the paraspinal muscle while still within the tolerable range of the patient. For the rRPMS control group, the stimulus intensity level will be set at 5% of the maximum output of the stimulator to minimize magnetic stimulation.
  Both groups will be exposed to an identical clicking sound generated during each session and the coil will be placed in contact with the patient (to have a similar sensation). The application of the rRPMS coil in both groups of patients will be conducted by experienced physiotherapists with sufficient preliminary training on the application of rPMS prior to the study.
  Arms: rPMS Intervention
Device: rPMS Controle — Both groups will undergo 10 sessions over a 2-week period. Each session will last 20 minutes and will be intermittent stimulation protocol consisting of 5 seconds of stimulation at a frequency of 20 Hz followed by 25 seconds of rest. The total number of stimulations over 20 minutes will be 4,000 pulses.
  The stimulation intensity level will be set at the level that induces sufficient contraction of the paraspinal muscle while still within the tolerable range of the patient. For the rRPMS control group, the stimulus intensity level will be set at 5% of the maximum output of the stimulator to minimize magnetic stimulation.
  Both groups will be exposed to an identical clicking sound generated during each session and the coil will be placed in contact with the patient (to have a similar sensation). The application of the rRPMS coil in both groups of patients will be conducted by experienced physiotherapists with sufficient preliminary training on the application of rPMS prior to the study.
  Arms: rPMS Controle

SUMMARY:
The aim of this study is to analyze the effect of Repeated Peripheral Magnetic Stimulation (rPMS) in patients with chronic low back pain. This is a controlled, randomized, multicenter clinical trial (Brazil x Portugal). The sample will consist of individuals with chronic low back pain with a score between 40 and 80 on the Oswestry scale, who will be randomly divided into 2 groups: control (CG) and intervention (IG). The instruments used for evaluation will be: visual analog pain scale (VAS), brief pain inventory (BPI), McGill questionnaire, Roland Morris scale and WHOQOL-BREF. Both groups will use the EMP device, with 10 sessions over a period of 2 weeks, in the IG applied in the flat tangential orientation lasting 20 minutes and an intermittent stimulation protocol consisting of 5 seconds of stimulation at a frequency of 20 Hz followed by 25 seconds of rest with a minimum intensity of 20% up to the maximum intensity to induce sufficient contraction of the paraspinal muscle and in the CG in transverse orientation with the stimulus intensity level set at 5% of the maximum output of the stimulator to minimize stimulation, both in the most painful lumbar region. The Wilcoxon test will be applied. Then, the Mann-Whitney test will be applied, adopting a significance level of 5%. It is expected that this research will contribute to more accurate protocols and evaluation methods for the EMP intervention, which generates responses in pain relief and non-surgical treatment.

DETAILED DESCRIPTION:
Low back pain is one of the most disabling and therapeutically challenging conditions affecting the population. Chronic low back pain is defined as pain and discomfort located below the rib margins and above the gluteal line, with or without pain referred to the lower limbs and represents a considerable challenge in terms of public health, with high financial costs. In Brazil, approximately 10 million Brazilians become disabled by this morbidity and at least 70% of the population will suffer an episode of low back pain in their lifetime.

In young adults, there are numerous studies on the impact of low back pain on functionality and therapeutic interventions, largely due to the high costs to the health service caused by the disability resulting from chronic low back pain in this economically active population. However, despite being identified as an important health problem, its consequences, as well as the effectiveness of therapeutic programs, are little known among the population.

Repetitive peripheral magnetic stimulation (rPMS) is a clinical treatment modality that depends on the generation of a powerful magnetic field by means of an electromagnetic coil. It is a low-intensity current capable of producing electrical impulses with variable frequencies of up to 200 Hz, thus being effective in the treatment of musculoskeletal pain, modeling and influencing pain neuroconduction processes. This electrical stimulation is capable of reducing pain through peripheral stimulation of large diameter fibers (A fibers), ending up inhibiting the entry of painful stimuli conducted by narrow diameter fibers (A delta and C fibers) closing the pain gate.

rPMS increases the cortical-motor excitability of the areas to be stimulated. This stimulation facilitates neuroplastic changes that improve motor recovery in the long term. Its beneficial effects on patients include increased muscle strength and mobility, decreased spasticity, analgesia, reduced edema, vasodilation, and decreased reflex inhibition, among others. However, to the best of our knowledge, no study has investigated the synergistic effects of SMP in patients with chronic low back pain with scores between 40 and 80 on the Oswestry scale. Therefore, it is extremely important to search for effective treatment modalities to improve pain and associated functional disability for the treatment of these patients.

OBJECTIVE General Objective To investigate the effects of rPMS treatment compared to a placebo treatment with the same equipment in reducing pain and functionality in patients with chronic low back pain.

Specific Objectives To verify whether rPMS alters the analgesic perception in the VAS, MPQ and BPI in patients with chronic low back pain; To verify whether rPMS alters the functionality of the lumbar spine by the ODI, RMDQ and WHOQOL-BREF in patients with chronic low back pain.

JUSTIFICATION Peripheral magnetic stimulation is a method indicated in the treatment of neuropathic pain syndromes, together with other forms of neurostimulation: electrical stimulation of the dorsal spine and deep brain stimulation. It is capable of bringing several benefits to patients, with an associated form of applicability and there are still few studies in patients with chronic low back pain, the application of this technique is justified to verify these effects in these patients. a modality.

METHODOLOGY Study design A controlled, randomized, multicenter clinical study will be conducted. Study location and population The study will be conducted at the Physiotherapy School Clinic of the Federal University of Alfenas (MG/Brazil), at the Neuroscience, Neuromodulation and Pain Study Laboratory - LANNED, located in the municipality of Alfenas, Minas Gerais, and at the Egas Moniz School of Health and Science (Portugal), at the Neuromodulation and Pain Unit - NeuroPain, in the municipality of Almada, Setúbal.

Sample Individuals with chronic low back pain with a score between 40 and 80 on the Oswestry scale will be selected, and 50 will be selected for treatment at the Physiotherapy School Clinic of the Federal University of Alfenas - MG and the Egas Moniz University Clinic - CUEM. The individuals will be divided into 2 groups: the control group and the intervention group.

Inclusion criteria The inclusion criteria considered: individuals with complaints of low back pain for more than three months, non-practitioners of sports activities, absence of significant spinal pathologies such as previous history of myelopathies, surgeries, instability or deformities in the spine (bone fractures), normal neurological examination for radiculopathies (patellar and Achilles tendon reflexes; voluntary motor function; sensitivity test).

Exclusion criteria The exclusion criteria are: trauma or systemic dysfunction; use of other alternative treatments; refusal to be randomized; protrusion or prolapse of one or more intervertebral discs with neurological symptoms; previous spinal surgery; infectious spondylopathy; low back pain secondary to inflammation, tumor or autoimmune disease; congenital spinal deformities; compression fracture caused by osteoporosis, spondylolysis or spondylolisthesis. Individuals who use prostheses; who have a history of seizures; have a history of epilepsy and have implanted or non-removable intracranial metal or devices.

Randomization of samples:

The volunteers will be divided into a control group and an intervention group through randomization. To do this, the participants will be allocated by another researcher, who will use the Research Randomizer website into two groups: Control Group (CG) and Intervention Group (IG).

Sample calculation The sample calculation performed estimates the number of 15 volunteers per group. This calculation will be performed to ensure a statistical power of 85% (β=0.20) and a significance level when p= 0.05.

Assessment Instruments:

Visual Analogue Scale (VAS) The VAS is a scale similar to a ruler, numbered with a starting point of zero and an ending point of ten, with 0 being no pain and 10 being the most unbearable pain felt at that moment by the patient.

The VAS was used to quantify the intensity and perception of the individual's pain, graded according to ordinal scores: no pain (0), mild pain (1 to 2), moderate (3 to 5) and severe (6 to 10).

Pressure Pain Threshold (PPT) PPTs will be assessed using a portable pressure algometer with a 1 cm2 rubber tip applicator and Bluetooth communication interface, placed perpendicularly on the skin with an application rate of 0 to 15 kgf/s (Physiocode brand). PPT will be defined as the minimum pressure first evoking a sensation of pain. PPTs will be measured twice with an interval of 10 seconds for each point, and the average value will be used for statistical analysis.

Algometry was used to examine the pain threshold for pressure applied between the spinous processes of the lumbar spine L1-L5.

McGill Pain Questionnaire (MPQ) The McGill Pain Questionnaire, also used to assess pain, is an instrument consisting of 78 descriptors (words that describe pain), organized into four categories (sensory, affective, evaluative, and mixed) and 20 subcategories. The individual is asked to choose one word from each subcategory, allowing the option of not choosing any. The analysis is performed by categories by adding the values associated with the chosen words and from the words selected by more than 30% of the population surveyed. Furthermore, this questionnaire is important for assessing pain from a multidimensional perspective, understanding that its development was based on the theoretical framework of pain physiology, which presupposes some universality of pain qualities and, finally, studies that confirmed that individuals with different sociocultural backgrounds, but with similar symptoms.

Brief Pain Inventory (BPI) Brief Pain Inventory - short form (Brief Pain Inventory - BPI): Multidimensional instrument that uses a scale of 0-10 to grade the following items: intensity, pain interference in the patient's ability to walk, daily activities, work, social activities, mood and sleep. The pain assessed by the patient is that experienced at the time of the questionnaire and the most intense, the least intense and the average pain of the last 24 hours.

Oswestry Scale (ODI) The Oswestry Scale (The Oswestry Disability Index, ODI) is a disease-specific instrument recommended for the assessment of spinal disorders. The ODI is an ordinal instrument, where 10 criteria are analyzed with six response alternatives for each criterion. The total score ranges from 0 to 100, with zero corresponding to normal function and 100 indicating great disability. For each item, zero is normality and five is the greatest functional alteration. The sum of the 10 questions divided by five multiplied by the number of questions answered, and multiplying everything by 100, constitutes the ODI.

Roland Morris Questionnaire (RMDQ) The Roland-Morris Brazil questionnaire (from the English and Roland Morris disability questionnaire, RMDQ) is specific to measure the functional disability of patients with low back pain, and consists of 24 questions related to activities of daily living, pain and function. For each affirmative question, 1 point is assigned. The score is the sum of the values, with a minimum score of "0" and a maximum score of "24". This questionnaire has a cut-off point of "14", that is, individuals evaluated with a score equal to or greater than "14" are classified as functionally disabled. Quality of life assessment instrument, abbreviated version (WHOQOL-BREF) The quality of life assessment instrument (WHOQOL-100) developed by the WHO Quality of Life Group in its abbreviated version (World Health Organization Quality of Life Bref, WHOQOL-BREF) will be used. This questionnaire consists of 26 questions (with questions 1 and 2 about general quality of life), and the answers follow a Likert scale (from 1 to 5, the higher the score, the better the quality of life). In addition to these two questions (1 and 2), the instrument has 24 facets that make up 4 domains: physical, psychological, social relationships and environment. Repeated Peripheral Magnetic Stimulation (rRPMS) Both groups will use the rRPMS device, with 10 sessions over a period of 2 weeks, in the IG applied in a flat tangential orientation lasting 20 minutes and an intermittent stimulation protocol consisting of 5 seconds of stimulation at a frequency of 20 Hz followed by 25 seconds of rest with a minimum intensity of 20% up to maximum intensity to induce sufficient contraction of the paraspinal muscle and in the CG in a transverse orientation with the stimulus intensity level set at 5% of the maximum output of the stimulator to minimize stimulation, both in the most painful lumbar region.

The group will be randomized into IG (n=25) and CG (n=25). It is known that a round coil is more advantageous than a figure-8 coil for stimulating structures in a deep layer such as spinal roots and covering a larger area such as a paravertebral muscle group. Thus, the investigators will use the round coil that will be more suitable for the treatment of low back pain.

The stimulation site will be determined based on the patient's most sensitive point before the start of each treatment session. For patients in the rPMS intervention group - in the prone position - the coil will be placed in a flat tangential orientation targeting the most painful lumbar region. This will allow the coil to be positioned parallel to the body surface, thus maximizing the effects of the magnetic stimulation applied to the area.

For patients in the rPMS control group, also in the prone position, the coil will be applied in a transverse orientation to the most painful lumbar region. This position of the coil, at a 90° angle to the body surface, will minimize the effects of magnetic stimulation applied to the area.

Both groups will undergo 10 sessions over a 2-week period. Each session will last 20 minutes and will use an intermittent stimulation protocol consisting of 5 seconds of stimulation at a frequency of 20 Hz followed by 25 seconds of rest. The total number of stimuli over 20 minutes will be 4,000 pulses.

The stimulation intensity level will be set at the level that induces sufficient contraction of the paraspinal muscle while still within the patient's tolerable range. For the rRPMS control group, the stimulus intensity level will be set at 5% of the maximum output of the stimulator to minimize magnetic stimulation.

Both groups will be exposed to an identical clicking sound generated during each session and the coil will be placed in contact with the patient (to have a similar sensation). The application of the rRPMS coil in both groups of patients will be conducted by experienced physiotherapists with sufficient preliminary training on the application of rPMS prior to the study.

Ethical Aspects

This project was submitted to the Ethics Committee of the Federal University of Alfenas for evaluation, and will comply with the precepts contained in resolution 466/12 of the National Health Council. It will also be submitted to the Egas Moniz Ethics Committee. Before starting to participate in this research, volunteers will receive all information related to the objectives and methodological procedures of the study and, after agreeing to participate, will sign the informed consent form. Participants will be informed about the objectives, research procedures, risks, benefits and minimization measures, and the data will be presented together. The informant may withdraw his/her participation at any time.

Statistical Procedures The Wilcoxon test will be used to assess possible differences between the results before and after the application of the treatment protocol in each group. The Mann-Whitney test will be used to assess the difference between the groups. A significance level of 0.05 will be adopted.

EXPECTED RESULTS It is expected that this research will contribute to more accurate protocols and evaluation methods for intervention with peripheral magnetic stimulation in chronic pain, as well as scientific basis for the technique.

RISKS AND BENEFITS:

The application of any therapeutic resource may expose the participant to some type of risk, however, this research is designed to minimize this occurrence as much as possible. Since it is an electromagnetic stimulation, the participant may feel some discomfort or pain, so he/she can end his/her participation immediately without any burden. It is expected that after the intervention of this research, it will bring benefits in improving chronic low back pain.

SANITARY MEASURES

Sanitary measures will be taken for both patients and researchers:

Exposure to sources of infection will be controlled, which is extremely important to protect patients and researchers and, thus, prevent outbreaks within the institution.

All health service professionals must wear face masks (surgical or N95/PFF2 or equivalent) for personal protection and source control (GVIMS/GGTES/ANVISA No. 07/2020); in addition, patients must wear the same mask.

Avoid close contact with people (i.e., maintain a distance of at least one meter), especially with those who have a fever, cough or sneezing; Practice respiratory etiquette (i.e., cover your mouth and nose with your forearm when coughing or sneezing with disposable tissues, discard them immediately after use in a closed trash can, and then sanitize your hands).

Wash your hands frequently with soap and water or with a 70% alcohol-based hand sanitizer and avoid touching your eyes, nose, and mouth with unwashed hands; It is known that viruses are inactivated by 70% alcohol and chlorine. Therefore, disinfect the surfaces of the location frequently.

ELIGIBILITY:
Inclusion Criteria:

Individuals with complaints of low back pain for more than three months

Non-practitioners of sports activities

Absence of significant spinal pathologies, such as previous history of myelopathies, surgeries, instabilities, or deformities (bone fractures)

Normal neurological examination for radiculopathies (patellar and Achilles tendon reflexes, voluntary motor function, and sensitivity test)

Exclusion Criteria:

Presence of trauma or systemic dysfunction

Use of other alternative treatments

Refusal to be randomized

Protrusion or prolapse of one or more intervertebral discs with neurological symptoms

Previous spinal surgery

Infectious spondylopathy

Low back pain secondary to inflammation, tumor, or autoimmune disease

Congenital spinal deformities

Compression fracture caused by osteoporosis, spondylolysis, or spondylolisthesis

Use of prosthesis

History of seizures or epilepsy

Implanted or non-removable intracranial metal or devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Change in chronic low back pain intensity measured by the Visual Analog Scale (VAS, 0-10; 0=no pain, 10=worst pain), categorized as no pain (0), mild (1-2), moderate (3-5), severe (6-10).

SECONDARY OUTCOMES:
Pressure Pain Threshold (L1-L5) | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Measures the pressure pain threshold (kgf/cm²) at lumbar levels L1-L5 using algometry; reflects local mechanical pain sensitivity.
McGill Pain Questionnaire (by category) | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Evaluates pain using sensory, affective, and evaluative descriptors, providing a qualitative profile of the pain experience.
Brief Pain Inventory - Intensity | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Subscale of the BPI (0-10) assessing average pain intensity during recent days.
Brief Pain Inventory - Interference | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Subscale of the BPI (0-10) measuring how pain interferes with daily activities, mood, sleep, and social relations.
Oswestry Disability Index (ODI) | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Disability index (0-100) related to low back pain; higher scores indicate greater functional limitation.
Roland-Morris Disability Questionnaire (RMDQ) | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Physical disability questionnaire (0-24) for low back pain; scores ≥14 indicate clinically significant limitation.
WHOQOL-BREF - Physical Domain | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Physical domain (1-5) of the WHOQOL-BREF assessing energy, mobility, and sleep.
WHOQOL-BREF - Psychological Domain | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Psychological domain (1-5) of the WHOQOL-BREF evaluating self-esteem, positive feelings, and thinking.
WHOQOL-BREF - Social Domain | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Social domain (1-5) of the WHOQOL-BREF covering personal relationships and social support.
WHOQOL-BREF - Environmental Domain | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions), and 4-week follow-up.
  Environmental domain (1-5) of the WHOQOL-BREF addressing safety, physical environment, and financial resources.
Treatment adherence (number of participants) | Assessments at baseline (Day 1), after 2 weeks (10 rPMS sessions)
  Number of participants who completed all 10 sessions of repetitive paravertebral magnetic stimulation (rPMS).

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health and Science, Almada, Setúbal District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD) from this study will not be shared due to ethical and privacy concerns. The collected information includes sensitive health data that, even if anonymized, could potentially lead to the identification of participants, especially given the relatively small sample size and the specific nature of the intervention. Furthermore, the informed consent obtained from participants does not include provisions for public data sharing.

REFERENCES:
- [Background] Lim YH, Song JM, Choi EH, Lee JW. Effects of Repetitive Peripheral Magnetic Stimulation on Patients With Acute Low Back Pain: A Pilot Study. Ann Rehabil Med. 2018 Apr;42(2):229-238. doi: 10.5535/arm.2018.42.2.229. Epub 2018 Apr 30. PMID 29765876
- [Background] Masse-Alarie H, Beaulieu LD, Preuss R, Schneider C. Repetitive peripheral magnetic neurostimulation of multifidus muscles combined with motor training influences spine motor control and chronic low back pain. Clin Neurophysiol. 2017 Mar;128(3):442-453. doi: 10.1016/j.clinph.2016.12.020. Epub 2016 Dec 28. PMID 28160750
- [Background] Diao Y, Pan J, Xie Y, Liao M, Wu D, Liu H, Liao L. Effect of Repetitive Peripheral Magnetic Stimulation on Patients With Low Back Pain: A Meta-analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2023 Sep;104(9):1526-1538. doi: 10.1016/j.apmr.2023.03.016. Epub 2023 Apr 26. PMID 37116558